CLINICAL TRIAL: NCT03815175
Title: XIENCE 28 USA Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10402
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Bleeding Disorder; Ischemic Stroke; Hemorrhagic Stroke; Hematological Diseases; Thrombocytopenia; Coagulation Disorder; Anemia; Renal Insufficiency; Coronary Artery Disease
Keywords: High Bleeding Risk (HBR); Dual antiplatelet therapy (DAPT); Drug eluting stent (DES); XIENCE; Percutaneous coronary intervention (PCI); Coronary Artery Disease
MeSH Terms: conditions — Hemostatic Disorders; Ischemic Stroke; Hemorrhagic Stroke; Hematologic Diseases; Thrombocytopenia; Anemia; Renal Insufficiency; Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- XIENCE (Experimental): XIENCE + 1 month DAPT
  Interventions: Device: XIENCE; Drug: DAPT (aspirin and/or P2Y12 receptor inhibitor)

INTERVENTIONS:
Device: XIENCE — Subjects who received XIENCE family stent systems will be included.
Drug: DAPT (aspirin and/or P2Y12 receptor inhibitor) — "1-month clear" subjects (pooled from Xience 28 USA study and Xience 28 Global study) will receive 1 month of DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days and will discontinue P2Y12 receptor inhibitor as early as 28 days and will continue with aspirin monotherapy through 12-month follow-up.
  Other Names: Dual antiplatelet therapy

SUMMARY:
The XIENCE 28 USA Study is prospective, single arm, multi-center, open label, non-randomized trial to evaluate safety of 1-month (as short as 28 days) dual antiplatelet therapy (DAPT) in subjects at high risk of bleeding (HBR) undergoing percutaneous coronary intervention (PCI) with the approved XIENCE family (XIENCE Xpedition Everolimus Eluting Coronary Stent System [EECSS], XIENCE Alpine EECSS and XIENCE Sierra EECSS) of coronary drug-eluting stents.

DETAILED DESCRIPTION:
The XIENCE 28 USA Study will evaluate the safety of 1-month DAPT following XIENCE implantation in HBR patients. A minimum of 640 to a maximum of 800 subjects will be registered from approximately 50 sites in the United States and Canada. Subject registration is capped at 75 per site. Eligibility of P2Y12 receptor inhibitor discontinuation will be assessed at 1-month follow-up. Subjects who are free from myocardial infarction (MI), repeat coronary revascularization, stroke, or stent thrombosis (ARC definite/probable) within 1 month (prior to 1-month visit but at least 28 days) after stenting AND have been compliant with 1-month DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days are considered as "1-month clear", and will discontinue P2Y12 receptor inhibitor as early as 28 days and continued with aspirin monotherapy through 12-month follow-up.

All registered subjects will be followed at 1, 3, 6 and 12 months post index procedure. The data collected from the XIENCE 28 USA Study will be pooled with the data from the XIENCE 28 Global Study (Protocol # ABT-CIP-10235) to compare with the historical control of non-complex HBR subjects treated with standard DAPT duration of up to 12 months from the XIENCE V USA Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is considered at high risk for bleeding (HBR), defined as meeting one or more of the following criteria at the time of registration and in the opinion of the referring physician, the risk of major bleeding with > 1-month DAPT outweighs the benefit:

   1. ≥ 75 years of age.
   2. Clinical indication for chronic (at least 6 months) or lifelong anticoagulation therapy
   3. History of major bleeding which required medical attention within 12 months of the index procedure.
   4. History of stroke (ischemic or hemorrhagic).
   5. Renal insufficiency (creatinine ≥ 2.0 mg/dl) or failure (dialysis dependent).
   6. Systemic conditions associated with an increased bleeding risk (e.g. hematological disorders, including a history of or current thrombocytopenia defined as a platelet count <100,000/mm3, or any known coagulation disorder associated with increased bleeding risk).
   7. Anemia with hemoglobin < 11g/dl.
2. Subject must be at least 18 years of age.
3. Subject must provide written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site prior to any trial related procedure.
4. Subject is willing to comply with all protocol requirements, including agreement to stop taking P2Y12 inhibitor at 1 month, if eligible per protocol.
5. Subject must agree not to participate in any other clinical trial for a period of one year following the index procedure, except for cases where subject is transferred to the XIENCE 90 study after the 1-month visit assessment

Angiographic Inclusion Criteria

1. Up to three target lesions with a maximum of two target lesions per epicardial vessel. Note:

   * The definition of epicardial vessels means left anterior descending coronary artery (LAD), left circumflex coronary artery (LCX) and right coronary artery (RCA) and their branches. For example, the subject must not have >2 lesions requiring treatment within both the LAD and a diagonal branch in total.
   * If there are two target lesions within the same epicardial vessel, the two target lesions must be at least 15 mm apart per visual estimation; otherwise this is considered as a single target lesion.
2. Target lesion must be located in a native coronary artery with visually estimated reference vessel diameter between 2.25 mm and 4.25 mm.
3. Exclusive use of XIENCE family of stent systems during the index procedure.
4. Target lesion has been treated successfully, which is defined as achievement of a final in-stent residual diameter stenosis of <20% with final TIMI-3 flow assessed by online quantitative angiography or visual estimation, with no residual dissection NHLBI grade ≥ type B, and no transient or sustained angiographic complications (e.g., distal embolization, side branch closure), no chest pain lasting > 5 minutes, and no ST segment elevation > 0.5mm or depression lasting > 5 minutes.

Exclusion Criteria:

1. Subject with an indication for the index procedure of acute ST-segment elevation MI (STEMI).
2. Subject has a known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, P2Y12 inhibitors (clopidogrel/prasugrel/ticagrelor), everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
3. Subject with implantation of another drug-eluting stent (other than XIENCE) within 12 months prior to index procedure.
4. Subject has a known left ventricular ejection fraction (LVEF) <30%.
5. Subject judged by physician as inappropriate for discontinuation from P2Y12 inhibitor use at 1 month, due to another condition requiring chronic P2Y12 inhibitor use.
6. Subject with planned surgery or procedure necessitating discontinuation of P2Y12 inhibitor within 1 month following index procedure.
7. Subject with a current medical condition with a life expectancy of less than 12 months.
8. Subject intends to participate in an investigational drug or device trial within 12 months following the index procedure. Transferring to the XIENCE 90 study will not be an exclusion criterion.
9. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
10. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
11. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.

Angiographic Exclusion Criteria

1. Target lesion is in a left main location.
2. Target lesion is located within an arterial or saphenous vein graft.
3. Target lesion is restenotic from a previous stent implantation.
4. Target lesion is a chronic total occlusion (CTO, defined as lesion with TIMI flow 0 for at least 3 months).
5. Target lesion is implanted with overlapping stents, whether planned or for bailout.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1605 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Mount Sinai Medical Center,New York, NY
Locations (111):
- United States (54):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - Scripps Memorial Hospital - La Jolla, La Jolla, California
  - Huntington Memorial Hospital, Pasadena, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Missouri Heart Center, Columbia, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Mount Sinai Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Joseph's Hospital Health Center, Syracuse, New York
  - Novant Health Heart and Vascular Research Institute, Charlotte, North Carolina
  - Cone Health Medical Group Heartcare, Greensboro, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - Kettering Medical Center, Kettering, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - UPMC Hamot, Erie, Pennsylvania
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Presbyterian Medical Center (PA), Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - Anmed Health, Anderson, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Heart Consultants, Knoxville, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor Scott and White Heart and Vascular Hospital, Dallas, Texas
  - Mission Research Institute, New Braunfels, Texas
  - HeartPlace Methodist Richardson, Richardson, Texas
  - East Texas Medical Center, Tyler, Texas
  - Mary Washington Hospital, Fredericksburg, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
- Kepler Universitätsklinikum GmbH, Linz, UPR AUS, Austria
- Belgium (4):
  - Onze-Lieve-Vrouwziekenhuis Campus Aalst, Aalst, Eflndrs
  - UZ Gent, Ghent, Flemish
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Jesse Ziekenhuis Campus Virga Jesse, Limbourg
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Saint John Regional Hospital - New Brunswick Heart Centre, Saint John, New Brunswick
  - Institute de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
  - Hopital du Sacre-Coeur de, Montreal, Quebec
- China (2):
  - Beijing AnZhen Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Jilin University, Changchun, N China
- Germany (7):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen, Bad-Wur
  - Elisabeth-Krankenhaus Essen GmbH, Essen, N. Rhin
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität MainzLangenbeckstrasse, Mainz, Rhinela
  - Herzzentrum Leipzig GmbH04289, Leipzig, Saxony
  - Segeberger Kliniken GmbH Am Kurpark 1, Bad Segeberg, Schlesw
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
  - UKE Hamburg (Universitatsklinik Eppendorf), Hamburg
- Hong Kong (3):
  - The University of Hong Kong (Queen Mary Hospital), Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
- Italy (8):
  - Clinica Mediterranea, Napoli, Campani
  - AOU Federico II - Università degli Studi di Napoli, Napoli, Campani
  - Az.Osp. Universitaria di Ferrara, Cona, Emi-rom
  - AOU di Parma, Parma, Emi-rom
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Rome, Lazio
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - Centro Cardiologico Monzino, Milan, Lombard
  - Istituto Clinico Humanitas, Rozzano, Lombard
- Netherlands (3):
  - Scheperziekenhuis Boermarkeweg, Emmen, Drenthe
  - Medisch Centrum Leeuwarden, Leeuwarden, Friesld
  - Albert Schweitzer Ziekenhuis Albert Schweitzerplaats, Dordrecht, Zuid
- Portugal (2):
  - Hospital de Santa Cruz, Carnaxide, Lisbon District
  - Santa Maria Hospital, Lisbon, Lisbon District
- Singapore (2):
  - National Heart Centre, Singapore, Central Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore Central
- Spain (7):
  - HCU Virgen de la Victoria Campus Universitario de Teatinos, Málaga, Andalu
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabr
  - Hospital del Mar Passeig Maritim de la Barceloneta, Barcelona, Catalon
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalon
  - Hospital Clinico Universitario de Valladolid, Valladolid, Cstleon
  - Hospital Alvaro Cunqueiro, Vigo, Pontev
  - Hospital Universitario Doce de Octubre, Madrid
- Switzerland (3):
  - Kantonsspital Aarau, Aarau, Basel
  - Center Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
- Taiwan (4):
  - Chang Gung Memorial Hospital, Linkou District, NTaiwan
  - National Taiwan University Hospital, Taipei, NTaiwan
  - Taipei Veterans General Hospital (VGH), Taipei, Ntaiwan
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, STailwan
- United Kingdom (6):
  - Freeman Hospital, High Heaton, Newcastle Upon Tyne
  - Craigavon Area Hospital, Portadown, Nirelnd
  - Southampton University Hospital, Southampton, Soeast
  - Royal Bournemouth Hospital, Bournemouth, Sowest
  - Royal Devon & Exeter Hospital, Exeter, Sowest
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Derived] Valgimigli M, Cao D, Angiolillo DJ, Bangalore S, Bhatt DL, Ge J, Hermiller J, Makkar RR, Neumann FJ, Saito S, Picon H, Toelg R, Maksoud A, Chehab BM, Choi JW, Campo G, De la Torre Hernandez JM, Kunadian V, Sardella G, Thiele H, Varenne O, Vranckx P, Windecker S, Zhou Y, Krucoff MW, Ruster K, Zheng Y, Mehran R; XIENCE 90 and XIENCE 28 Investigators. Duration of Dual Antiplatelet Therapy for Patients at High Bleeding Risk Undergoing PCI. J Am Coll Cardiol. 2021 Nov 23;78(21):2060-2072. doi: 10.1016/j.jacc.2021.08.074. PMID 34794687
- [Derived] Valgimigli M, Cao D, Makkar RR, Bangalore S, Bhatt DL, Angiolillo DJ, Saito S, Ge J, Neumann FJ, Hermiller J, Picon H, Toelg R, Maksoud A, Chehab BM, Wang LJ, Wang J, Mehran R. Design and rationale of the XIENCE short DAPT clinical program: An assessment of the safety of 3-month and 1-month DAPT in patients at high bleeding risk undergoing PCI with an everolimus-eluting stent. Am Heart J. 2021 Jan;231:147-156. doi: 10.1016/j.ahj.2020.09.019. Epub 2020 Oct 6. PMID 33031789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1605 subjects were enrolled in XIENCE 28 study. The XIENCE 28 USA study was conducted at 58 sites in the US and Canada between February 25, 2019 and February 7, 2020. While XIENCE 28 Global study was conducted at 52 sites in Europe and Asia between February 9, 2018 and April 22, 2019.
Pre-assignment Details: The data collected from the XIENCE 28 USA Study was pooled with the data from the XIENCE 28 Global Study (NCT # NCT03355742) to compare with the historical control of non-complex HBR subjects treated with standard DAPT duration of up to 12 months from the XIENCE V USA Study.
Groups:
- XIENCE: XIENCE + 1 month dual antiplatelet therapy (DAPT)
  XIENCE: Subjects who received XIENCE family stent systems will be included.
  DAPT (aspirin and/or P2Y12 receptor inhibitor): "1-month clear" subjects (pooled from Xience 28 USA study and Xience 28 Global study) will receive 1 month of DAPT without interruption of either aspirin and/or P2Y12 receptor inhibitor for > 7 consecutive days and will discontinue P2Y12 receptor inhibitor as early as 28 days and will continue with aspirin monotherapy through 12-month follow-up.
Period: Overall Study
Arm/Group | XIENCE
Started | 1605
Completed | 1439
Not Completed | 166
Not completed — Subject Lost to Follow-up | 6
Not completed — Subject Withdrew Consent | 48
Not completed — Subject Withdrawn by Physician/Site | 10
Not completed — Death | 86
Not completed — Improper/Duplicate SubjectEnrollment | 1
Not completed — Subject Discontinued by Sponsor | 2
Not completed — Other Status Change Reason | 1
Not completed — Missed Visit | 12

BASELINE CHARACTERISTICS:
Arm/Group | XIENCE
Number analyzed (Participants) | 1605
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.15 (8.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 538
  Male | 1067
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 137
  Black or African American | 42
  Hispanic or Latino | 168
  Native Hawaiian or Pacific Islander | 0
  White | 939
  Did Not Wish to Disclose | 40
  Not Available | 445
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 327
  Italy | 231
  Canada | 70
  United States | 572
  Hong Kong | 48
  Belgium | 64
  Spain | 89
  Netherlands | 49
  Switzerland | 37
  Taiwan | 48
  Singapore | 22
  United Kingdom | 30
  China | 7
  Portugal | 8
  Austria | 3
Prior Percutaneous Coronary Intervention (PCI) [Count of Participants; unit: Participants] | 451

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Rate of All Death or All Myocardial Infarction (MI) (Modified Academic Research Consortium [ARC]), by Propensity Score Quintile
Description: All death: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g.cancer, infection) should be classified as cardiac.
  MI Definition (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Peripheral MI
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
percentage of participants
  Adjusted Overall Rate | 3.5
  Q1: number analyzed (Participants) | 46
  Q1 | 4.3
  Q2: number analyzed (Participants) | 148
  Q2 | 4.1
  Q3: number analyzed (Participants) | 266
  Q3 | 2.6
  Q4: number analyzed (Participants) | 407
  Q4 | 2.7
  Q5: number analyzed (Participants) | 513
  Q5 | 3.9
Statistical Analysis 1: Comparison: XIENCE; Test type: Non-Inferiority — H0: Death/(MI[1m-DAPT]) - Death/(MI [XIENCE V USA]) ≥ δ HA: Death/MI([1m-DAPT]) - Death/(MI [XIENCE V USA: NCT00676520]) < δ Where δ is the non-inferiority margin. The test will be carried out with a one-sided significance level of 0.025 and a non-inferiority margin (δ) of 2.5%; p = 0.0005, Farrington-Manning method

2. Primary Outcome: Percentage of Participants With Composite Rate of All Death or All Myocardial Infarction (Modified ARC), by Propensity Score Quintile
Description: as for outcome 1
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
percentage of participants
  Adjusted Overall Rate | 3.2
  Q1: number analyzed (Participants) | 46
  Q1 | 0.0
  Q2: number analyzed (Participants) | 146
  Q2 | 2.7
  Q3: number analyzed (Participants) | 263
  Q3 | 3.4
  Q4: number analyzed (Participants) | 401
  Q4 | 5.5
  Q5: number analyzed (Participants) | 500
  Q5 | 4.4

3. Primary Outcome: Percentage of Participants With Composite Rate of All Death or All Myocardial Infarction (Modified ARC), by Propensity Score Quintile
Description: as for outcome 1
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
percentage of participants
  Adjusted Overall Rate | 6.7
  Q1: number analyzed (Participants) | 46
  Q1 | 4.3
  Q2: number analyzed (Participants) | 149
  Q2 | 6.7
  Q3: number analyzed (Participants) | 267
  Q3 | 6.0
  Q4: number analyzed (Participants) | 406
  Q4 | 7.9
  Q5: number analyzed (Participants) | 513
  Q5 | 8.4

4. Secondary Outcome: Percentage of Participants With Major Bleeding Rate (Bleeding Academic Research Consortium [BARC] Type 2-5), by Propensity Score Quintiles
Description: Bleeding per Bleeding Academic Research Consortium (BARC) adjudicated definitions:
  * Type 2: Any overt, actionable sign of hemorrhage
  * Type 3a: Overt bleeding plus Hb drop of 3 to < 5g/dL;Any transfusion with overt bleeding
  * Type 3b: Overt bleeding plus Hb drop ≥ 5 g/dL;Cardiac tamponade;Bleeding requiring surgical intervention for control;Bleeding requiring IV vasoactive agents
  * Type 3c: Intracranial hemorrhage; Subcategories confirmed by autopsy/imaging/lumbar puncture;Intraocular bleed compromising vision
  * Type 4: CABG-related bleeding: Perioperative intracranial bleeding within 48h;Reoperation after closure of sternotomy for the purpose of controlling bleeding;Transfusion of ≥ 5 U whole blood/packed red blood cells within a 48h period;Chest tube output ≥ 2L within 24-h period
  * Type 5: Fatal bleeding
  * Type 5a: Probable fatal bleeding;no autopsy/imaging confirmation but clinically suspicious
  * Type 5b: Definite fatal bleeding;overt bleeding/autopsy/imaging confirmation
Time Frame: From 1 to 6 months
Population: The number of participants analyzed for each time frame and outcome measure will vary based on:
  1. Number of subjects who actually completed follow-up for the given time point analyzed
  2. The denominator rule used to calculate event rates: subjects that were lost to follow-up, or withdrew consent, or died before the time point of interest, without having the endpoint of interest are excluded from the denominator.
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1362
percentage of participants
  Adjusted Overall Rate | 4.9
  Q1: number analyzed (Participants) | 46
  Q1 | 4.3
  Q2: number analyzed (Participants) | 146
  Q2 | 5.5
  Q3: number analyzed (Participants) | 263
  Q3 | 2.3
  Q4: number analyzed (Participants) | 404
  Q4 | 5.2
  Q5: number analyzed (Participants) | 503
  Q5 | 7.0
Statistical Analysis 1: Comparison: XIENCE; Test type: Superiority — H0: B (1m-DAPT) - B (XIENCE V USA) ≥ 0 HA: B (1m-DAPT) - B (XIENCE V USA: NCT00676520) < 0 B 1m-DAPT and B XIENCE V USA are bleeding rates (BARC type 2-5) between 1-month and 6-month follow-up for the pooled 1-month DAPT arm and XIENCE V USA historical control, respectively; p = 0.1888, Farrington and Manning method

5. Secondary Outcome: Percentage of Participants With Major Bleeding Rate (BARC Type 2-5), by Propensity Score Quintiles
Description: as for outcome 4
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1325
percentage of participants
  Adjusted Overall Rate | 2.5
  Q1: number analyzed (Participants) | 46
  Q1 | 2.2
  Q2: number analyzed (Participants) | 145
  Q2 | 1.4
  Q3: number analyzed (Participants) | 257
  Q3 | 3.1
  Q4: number analyzed (Participants) | 392
  Q4 | 2.0
  Q5: number analyzed (Participants) | 485
  Q5 | 3.7

6. Secondary Outcome: Percentage of Participants With Major Bleeding Rate (BARC Type 2-5), by Propensity Score Quintiles
Description: as for outcome 4
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1333
percentage of participants
  Adjusted Overall Rate | 7.1
  Q1: number analyzed (Participants) | 46
  Q1 | 6.5
  Q2: number analyzed (Participants) | 146
  Q2 | 6.8
  Q3: number analyzed (Participants) | 259
  Q3 | 5.4
  Q4: number analyzed (Participants) | 395
  Q4 | 6.8
  Q5: number analyzed (Participants) | 487
  Q5 | 10.1

7. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: Definite stent thrombosis:
  Definite stent thrombosis is considered to have occurred by either angiographic or pathologic confirmation.
  Probable stent thrombosis:
  Clinical definition of probable stent thrombosis is considered to have occurred after intracoronary stenting in the following cases:
  * Any unexplained death within the first 30 days
  * Irrespective of the time after the index procedure, any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause
Time Frame: From 1 to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1361
Participants | 4

8. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: as for outcome 7
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1328
Participants | 0

9. Secondary Outcome: Number of Participants With Stent Thrombosis (ARC Definite/Probable, ARC Definite)
Description: as for outcome 7
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1333
Participants | 4

10. Secondary Outcome: Number of All Death (Cardiac Death, Vascular Death, Non-cardiovascular Death)
Description: All Death:
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even inpatients with coexisting potentially fatal non-cardiac disease (e.g. cancer,infection) should be classified as cardiac.
  Cardiac death:
  Any death due to proximate cardiac cause (e.g. MI, low-output failure,fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death:
  Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death:
  Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 23

11. Secondary Outcome: Number of All Death (Cardiac Death, Vascular Death, Non-cardiovascular Death)
Description: as for outcome 10
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 40

12. Secondary Outcome: Number of All Death (Cardiac Death, Vascular Death, Non-cardiovascular Death)
Description: as for outcome 10
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 64

13. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI) and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: All Myocardial Infarction (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URL with baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
  TV-MI: All infarcts that cannot be clearly attributed to a vessel other than the target vessel will be considered related to the target vessel.
Time Frame: From 1 to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 24

14. Secondary Outcome: Number of Participants With All MI and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: as for outcome 13
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 18

15. Secondary Outcome: Number of Participants With All MI and MI Attributed to Target Vessel (TV-MI, Modified ARC)
Description: as for outcome 13
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 41

16. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: Cardiac death:
  Any death due to proximate cardiac cause (e.g. MI, low-output failure,fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI:
    * Within 48h after PCI: CK-MB >3 x URL or Troponin > 3 x URLwith baseline value < URL
    * Within 72h after CABG: CK-MB >5 x URL or Troponin > 5 x URL with baseline value < URL
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 35

17. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: as for outcome 16
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 33

18. Secondary Outcome: Number of Participants With Composite of Cardiac Death or MI (Modified ARC)
Description: as for outcome 16
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 68

19. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: All death: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g.cancer, infection) should be classified as cardiac.
  MI (Modified ARC):
  Patients present any of the following clinical or imaging evidence of ischemia:
  * Clinical symptoms of ischemia;
  * ECG changes indicative of new ischemia - new ST-T changes or new left bundle branch block (LBBB), development of pathological Q waves;
  * Imaging evidence of a new loss of viable myocardium or a new regional wall motion abnormality)
  AND confirmed with elevated cardiac biomarkers per ARC criteria:
  * Periprocedural MI
  * Spontaneous MI (> 48h following PCI, > 72h following CABG): CK-MB > URL or Troponin > URL with baseline value < URL
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 46

20. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: as for outcome 19
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 57

21. Secondary Outcome: Number of Participants With Composite of All Death or All MI (Modified ARC)
Description: as for outcome 19
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 103

22. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke and Hemorrhagic Stroke)
Description: An acute symptomatic episode of neurological dysfunction attributed to a vascular cause lasting more than 24 hours or lasting 24 hours or less with a brain imaging study or autopsy showing new infarction.
  * Ischemic Stroke: An acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of central nervous system tissue.
  * Hemorrhagic Stroke: An acute symptomatic episode of focal or global cerebral or spinal dysfunction caused by a non-traumatic intraparenchymal, intraventricular, or subarachnoid hemorrhage.
  * Undetermined Stroke: A stroke with insufficient information to allow categorization as ischemic or hemorrhagic.
  * Pharmacologic, i.e., thrombolytic drug administration, or Non-pharmacologic, i.e., neurointerventional procedure (e.g., intracranial angioplasty)
Time Frame: From 1 to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1357
Participants | 4

23. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke and Hemorrhagic Stroke)
Description: as for outcome 22
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1320
Participants | 7

24. Secondary Outcome: Number of Participants With All Stroke (Ischemic Stroke and Hemorrhagic Stroke)
Description: as for outcome 22
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1321
Participants | 11

25. Secondary Outcome: Number of Participants With Clinically-indicated Target Lesion Revascularization (CI-TLR)
Description: Target Lesion Revascularization (TLR) is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography.
  Clinically Indicated [CI] Revascularization:
  A revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test
  * A TLR/TVR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 10

26. Secondary Outcome: Number of Participants With CI-TLR
Description: as for outcome 25
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 8

27. Secondary Outcome: Number of Participants With CI-TLR
Description: as for outcome 25
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 18

28. Secondary Outcome: Number of Participants With Clinically-indicated Target Vessel Revascularization (CI-TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
  A revascularization is considered clinically indicated if angiography at follow-up shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  * A positive history of recurrent angina pectoris, presumably related to the target vessel;
  * Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  * Abnormal results of any invasive functional diagnostic test (e.g.,Doppler flow velocity reserve, fractional flow reserve);
  * A TVR with a diameter stenosis ≥70% in the absence of the above mentioned ischemic signs or symptoms.
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 14

29. Secondary Outcome: Number of Participants With CI-TVR
Description: as for outcome 28
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 15

30. Secondary Outcome: Number of Participants With CI-TVR
Description: as for outcome 28
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 29

31. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: TLF is defined as a composite of all cardiac death, myocardial infarction attributed to target vessel or clinically-indicated TLR.
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 35

32. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: as for outcome 31
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 34

33. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF, Composite of Cardiac Death, TV-MI and CI-TLR)
Description: as for outcome 31
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 69

34. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, Composite of Cardiac Death, TV-MI and CI-TVR)
Description: TVF is defined as a composite of cardiac death, MI attributed to target vessel, clinically-indicated TLR, or clinically-indicated TVR, non-TLR.
Time Frame: From 1 to 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1380
Participants | 38

35. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, Composite of Cardiac Death, TV-MI and CI-TVR)
Description: as for outcome 34
Time Frame: From 6 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1356
Participants | 39

36. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF, Composite of Cardiac Death, TV-MI and CI-TVR)
Description: as for outcome 34
Time Frame: From 1 to 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1381
Participants | 77

37. Secondary Outcome: Number of Participants With Major Bleeding Defined by the Bleeding Academic Research Consortium (BARC) Type 3-5
Description: Bleeding per Bleeding Academic Research Consortium (BARC) adjudicated definitions are as follows:
  * Type 3a: Overt bleeding plus Hemoglobin(Hb) drop of 3 to < 5 g/dL; Any transfusion with overt bleeding
  * Type 3b: Overt bleeding plus Hb drop ≥ 5 g/dL; Cardiac tamponade; Bleeding requiring surgical intervention for control; Bleeding requiring IV vasoactive agents
  * Type 3c: Intracranial hemorrhage;Subcategories confirmed by autopsy or imaging or lumbar puncture; Intraocular bleed compromising vision
  * Type 4: CABG-related bleeding: Perioperative intracranial bleeding within 48 h; Reoperation after closure of sternotomy for the purpose of controlling bleeding; Transfusion of ≥ 5 U whole blood or packed red blood cells within a 48-h period; Chest tube output ≥ 2L within a 24-h period
  * Type 5: Fatal bleeding
  * Type 5a: Probable fatal bleeding; no autopsy/imaging confirmation but clinically suspicious
  * Type 5b: Definite fatal bleeding;overt bleeding/autopsy or imaging confirmation
Time Frame: From 1 to 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1362
Participants | 33

38. Secondary Outcome: Number of Participants With Major Bleeding Defined by the Bleeding Academic Research Consortium (BARC) Type 3-5
Description: as for outcome 37
Time Frame: From 6 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1325
Participants | 18

39. Secondary Outcome: Number of Participants With Major Bleeding Defined by the Bleeding Academic Research Consortium (BARC) Type 3-5
Description: as for outcome 37
Time Frame: From 1 to 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | XIENCE
Number analyzed (Participants) | 1333
Participants | 49

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | XIENCE
All-Cause Mortality (participants affected / at risk) | 86/1605
Serious Adverse Events (participants affected / at risk) | 615/1605
Other Adverse Events (participants affected / at risk) | 296/1605
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE (N=1605)
Anaemia (Blood and lymphatic system disorders) | 18
Bicytopenia (Blood and lymphatic system disorders) | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 4
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 91
Angina Unstable (Cardiac disorders) | 1
Aortic Valve Incompetence (Cardiac disorders) | 3
Aortic Valve Stenosis (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 49
Atrial Flutter (Cardiac disorders) | 5
Atrial Tachycardia (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 2
Atrioventricular Block Complete (Cardiac disorders) | 5
Atrioventricular Block Second Degree (Cardiac disorders) | 1
Bifascicular Block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 6
Cardiac Arrest (Cardiac disorders) | 3
Cardiac Failure (Cardiac disorders) | 32
Cardiac Failure Acute (Cardiac disorders) | 8
Cardiac Failure Chronic (Cardiac disorders) | 4
Cardiac Failure Congestive (Cardiac disorders) | 34
Cardiac Tamponade (Cardiac disorders) | 1
Cardiogenic Shock (Cardiac disorders) | 3
Cardiomegaly (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 2
Congestive Cardiomyopathy (Cardiac disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 9
Coronary Artery Stenosis (Cardiac disorders) | 2
Diastolic Dysfunction (Cardiac disorders) | 1
Dressler's Syndrome (Cardiac disorders) | 1
Ischaemic Cardiomyopathy (Cardiac disorders) | 1
Mitral Valve Incompetence (Cardiac disorders) | 6
Myocardial Infarction (Cardiac disorders) | 30
Myocardial Ischaemia (Cardiac disorders) | 2
Myopericarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pleuropericarditis (Cardiac disorders) | 1
Pulseless Electrical Activity (Cardiac disorders) | 1
Right Ventricular Failure (Cardiac disorders) | 2
Sick Sinus Syndrome (Cardiac disorders) | 4
Sinoatrial Block (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 2
Supraventricular Tachycardia (Cardiac disorders) | 3
Tachyarrhythmia (Cardiac disorders) | 4
Tachycardia (Cardiac disorders) | 1
Tricuspid Valve Incompetence (Cardiac disorders) | 2
Ventricular Extrasystoles (Cardiac disorders) | 4
Ventricular Fibrillation (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 6
Vertigo (Ear and labyrinth disorders) | 3
Vertigo Positional (Ear and labyrinth disorders) | 2
Hyperparathyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Retinal Artery Occlusion (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 3
Colitis Ulcerative (Gastrointestinal disorders) | 1
Colonic Polyp (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Duodenal Ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 3
Faeces Discoloured (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastritis Erosive (Gastrointestinal disorders) | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Inguinal Hernia (Gastrointestinal disorders) | 2
Intestinal Ischaemia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Pancreatitis Necrotising (Gastrointestinal disorders) | 1
Rectal Ulcer (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2
Varices Oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Catheter Site Haemorrhage (General disorders) | 1
Chest Discomfort (General disorders) | 2
Chest Pain (General disorders) | 9
Death (General disorders) | 23
Dysplasia (General disorders) | 1
Fatigue (General disorders) | 1
General Physical Health Deterioration (General disorders) | 1
Hernia Obstructive (General disorders) | 1
Impaired Healing (General disorders) | 1
Multi-Organ Failure (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 3
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 3
Cholangitis (Hepatobiliary disorders) | 4
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis Acute (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic Cirrhosis (Hepatobiliary disorders) | 2
Jaundice Cholestatic (Hepatobiliary disorders) | 1
Abdominal Infection (Infections and infestations) | 1
Abscess Limb (Infections and infestations) | 2
Arthritis Infective (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Cholecystitis Infective (Infections and infestations) | 1
Corona Virus Infection (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 3
Endocarditis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Gallbladder Abscess (Infections and infestations) | 1
Gangrene (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 5
Haematoma Infection (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 4
Infectious Pleural Effusion (Infections and infestations) | 1
Influenza (Infections and infestations) | 3
Lobar Pneumonia (Infections and infestations) | 2
Localised Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Lung Abscess (Infections and infestations) | 1
Muscle Abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis Externa (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 36
Postoperative Wound Infection (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 6
Sepsis (Infections and infestations) | 14
Sepsis Syndrome (Infections and infestations) | 2
Septic Shock (Infections and infestations) | 7
Severe Acute Respiratory Syndrome (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Soft Tissue Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 17
Urosepsis (Infections and infestations) | 3
Vulval Abscess (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 3
Clavicle Fracture (Injury, poisoning and procedural complications) | 1
Compression Fracture (Injury, poisoning and procedural complications) | 1
Cranial Nerve Injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 8
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 6
Foot Fracture (Injury, poisoning and procedural complications) | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Patella Fracture (Injury, poisoning and procedural complications) | 3
Pelvic Fracture (Injury, poisoning and procedural complications) | 2
Perirenal Haematoma (Injury, poisoning and procedural complications) | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 2
Tibia Fracture (Injury, poisoning and procedural complications) | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 5
Wound Dehiscence (Injury, poisoning and procedural complications) | 1
Arteriogram Coronary (Investigations) | 1
Blood Glucose Increased (Investigations) | 1
Blood Pressure Abnormal (Investigations) | 1
Blood Pressure Increased (Investigations) | 1
Blood Urine Present (Investigations) | 1
Cardiac Stress Test Abnormal (Investigations) | 1
Ejection Fraction Decreased (Investigations) | 1
Electrocardiogram Abnormal (Investigations) | 1
Heart Rate Decreased (Investigations) | 1
Hepatic Enzyme Increased (Investigations) | 1
Troponin Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 3
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2
Fluid Overload (Metabolism and nutrition disorders) | 7
Gout (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Fistula (Musculoskeletal and connective tissue disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1
Acute Lymphocytic Leukaemia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Biliary Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal Tract Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases To Central Nervous (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleural Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Carotid Artery Disease (Nervous system disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 2
Cauda Equina Syndrome (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 15
Cognitive Disorder (Nervous system disorders) | 2
Complex Regional Pain Syndrome (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Dizziness Postural (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hepatic Encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Loss Of Consciousness (Nervous system disorders) | 1
Lumbar Radiculopathy (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 2
Neurodegenerative Disorder (Nervous system disorders) | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 15
Transient Ischaemic Attack (Nervous system disorders) | 5
Viith Nerve Paralysis (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Mental Disorder (Psychiatric disorders) | 1
Diabetic Nephropathy (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 3
Prerenal Failure (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 7
Renal Failure Acute (Renal and urinary disorders) | 20
Renal Failure Chronic (Renal and urinary disorders) | 6
Urinary Retention (Renal and urinary disorders) | 2
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 3
Prostatomegaly (Reproductive system and breast disorders) | 1
Scrotal Mass (Reproductive system and breast disorders) | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5
Angioedema (Skin and subcutaneous tissue disorders) | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 4
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 1
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1
Cataract Operation (Surgical and medical procedures) | 1
Colon Polypectomy (Surgical and medical procedures) | 1
Hip Arthroplasty (Surgical and medical procedures) | 1
Hospitalisation (Surgical and medical procedures) | 1
Limb Immobilisation (Surgical and medical procedures) | 1
Mitral Valve Repair (Surgical and medical procedures) | 1
Osteomyelitis Drainage (Surgical and medical procedures) | 1
Aortic Stenosis (Vascular disorders) | 10
Arteriovenous Fistula (Vascular disorders) | 2
Deep Vein Thrombosis (Vascular disorders) | 3
Femoral Arterial Stenosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 84
Hypertension (Vascular disorders) | 2
Hypertensive Crisis (Vascular disorders) | 8
Hypertensive Emergency (Vascular disorders) | 2
Hypotension (Vascular disorders) | 5
Intermittent Claudication (Vascular disorders) | 1
Orthostatic Hypotension (Vascular disorders) | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 3
Peripheral Ischaemia (Vascular disorders) | 4
Peripheral Vascular Disorder (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vascular Stenosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE (N=1605)
Angina Pectoris (Cardiac disorders) | 123
Haemorrhage (Vascular disorders) | 173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT03815175/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT03815175/SAP_001.pdf